CLINICAL TRIAL: NCT04372966
Title: Prospective, Double Blind Randomised Controlled Trial Comparing the Uncemented (CORAIL, DePuy) Versus Cemented (Exeter) Total Knee Arthroplasty for Displaced Subcapital Hip Fractures
Brief Title: Uncemented Versus Cemented Total Hip Arthroplasty for Displaced Intracapsular Hip Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Chief Investigator (John Keating)
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06/S0501/80
Record Dates: First submitted 2020-04-27; First posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Intervention Model Description: Randomaised controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cemented (Active Comparator): This group will receive a cemented Exeter stem and contemporary acetabular component (Stryker).
  Interventions: Device: Total hip arthroplasty
- Uncemented (Active Comparator): This group will receive an uncemented Corail stem and uncemented acetabular component (Depuy).
  Interventions: Device: Total hip arthroplasty

INTERVENTIONS:
Device: Total hip arthroplasty — Corail Total hip arthroplasty system, Depuy. Exeter and Contemporary acetabular components, Stryker.
  Other Names: Total hip replacement

SUMMARY:
Displaced subcapital hip fractures are very common and account for almost 50% of all hip fractures. The aim of the present study is to determine whether an uncemented total hip replacement is better than conventional cemented hip replacement to treat these fractures.

DETAILED DESCRIPTION:
Hip fractures account for 20% of all fractures and displaced subcapital fractures represent 45% of the hip fracture workload. All of these patients are treated with some form of hip replacement. Recent randomised trials have confirmed that total hip replacement is probably the best choice of treatment in a fit older patient and is better than partial hip replacement or repair of the fracture with screws which are the other most commonly used treatments. Hip replacements may be cemented or uncemented. The uncemented type of hip replacement has not been commonly used in this group of patients but may have some advantages. The uncemented hip replacement is a shorter operation and this may be advantageous in the hip fracture population group since these are older patients, many of whom have other medical problems. The use of cement is occasionally associated with development of heart problems during anaesthesia.

Participants: The original aim was to recruit 200 patients who have been admitted with a displaced subcapital hip fracture to the New Royal Infirmary and will undergo total hip replacement surgery within 48 hours of admission. Patients fitting the inclusion criteria will be given a patient information sheet and will be given between 24-48 hours to decide whether they give consent to participate in the trial. Patients who have given their consent will be randomly allocated to one of two groups i.e.. allocation to one of the two groups will entirely by chance. Each group will have 100 patients.

Intervention Both groups will received a total hip replacement. The only difference between the two groups is the type of hip replacement and the way it is fixed in the thigh bone. One type of hip replacement requires cement ('Exeter'), the other ('CORAIL' from DePuy) doesn't. Other surgical protocols and care after the surgery will be exactly the same for both groups.

Purpose The purpose of this research is to compare the clinical outcome (i.e. complications, revisions etc.) and the function of the patients between the two groups at several different time points: around 8 weeks, 4 months, 12 months and 24 months post surgery.

Outcome measures Clinical: Surgery complications, duration of surgery, readmissions, revision surgery, duration of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* patients over the age of 60 years with a displaced intracapsular hip fracture and are admitted to the study centre and are under the care of four orthopaedic trauma surgeons
* patients who were independently mobile before their hip fracture
* patients without cognitive impairment (mini-mental score >6) and able to give informed consent
* patients without serious concomitant disease

Exclusion Criteria:

* those not meeting the inclusion criteria
* patients who are not independently mobile outside the home
* unable to give informed consent
* serious concomitant disease with anaesthetic risk too great for Tsurgery

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-09-24 (Actual); Primary Completion 2011-12-29 (Actual); Study Completion 2016-12-29 (Actual)

PRIMARY OUTCOMES:
Hip specific function | 1 year
  This was measured using the Oxford hip score which ranges from 0 (worst score) to 48 (best score) points.

SECONDARY OUTCOMES:
Hip specific function | 6 and 72 months
  Oxford hip score which ranges from 0 (worst score) to 48 (best score) points.
Hip specific function | 6, 12 and 72 months
  Harris Hip Score which ranges from 0 (worst score) to 100 (best score) points.
Generic health | 6, 12 and 72 months
  Euro Qol 5-dimension scale (3L) which ranges from -0.594 to 1, where 1 represents perfect health and 0 represents death. Negative values represent a state perceived as worse than death.
Mobility | 6 months
  Timed get up and go test
Subjective patient hip pain | 6, 12 and 72 months
  Pain visual analogue scale from 1 (no pain) to 10 (maximum pain)
Operative time | At time of index surgery
  Time from knife to skin to wound closure
Intraoperative blood loss | At time of of surgery
  Amount of blood lost during the index proceedure
Patient satisfaction | 6, 12 and 72 months
  Overall how satisfied are you with the results of your hip replacement surgery?" The response to each question was recorded using a five-point Likert scale: very satisfied, somewhat satisfied, neutral, somewhat dissatisfied, and very dissatisfied.
Complications | Time of surgery until one year following surgery
  Rate of complications (intra / post operative)
Survival | Time of index surgery until final follow up (72 months), revision or death
  Kaplan Meier assessment of implant survival

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Lothian, Edinburgh, Edinburgh City, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This is not planned